CLINICAL TRIAL: NCT00838994
Title: A Randomized Controlled Trial of Acupuncture for Residual Insomnia Associated With Major Depressive Disorder
Brief Title: Acupuncture for Residual Insomnia Associated With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Baptist University (Other)
Responsible Party: Dr. Chung Ka-Fai/ Associate Professor, Department of Psychiatry, the University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACUP-002
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Electroacupuncture; Acupuncture; Randomized Clinical Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional Acupuncture (Experimental): Patients will be treated at bilateral Ear Shenmen, Sishencong EX-HN1, Anmian, and unilateral Yintang EX-HN3 and Baihui GV20. Acupuncture treatment will be performed by a registered Chinese medicine practitioner. "De qi"(an irradiating feeling considered to be indicative of effective needling) is achieved if possible. An electric-stimulator (CEFAR Acus II, Lund, Sweden) is connected to these needles to give an electric-stimulation in continuous wave, frequency of 4 Hz, 0.45 ms square wave pulses and constant current. Surgical tape or hair pin will be adhered to the needles.The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Interventions: Other: Acupuncture
- Minimal Acupuncture (Active Comparator): Patients will be treated superficially at points away from classic acupoints. The points include bilateral "Deltoideus" [in the middle of the line insertion of Binao LI 14 and acromion], "Forearm" [1 inch laterally of the middle point between Shaohai HE3 and Shenmen HE7], "Upper arm" [1 inch laterally of Tianfu LU 3] and "Lower leg" [0.5 inch dorsally of Xuanzhong GB39]. "De qi" is avoided during needling. The treatment procedure, electric-stimulation, frequency, duration and number of treatment sessions will be the same for the Traditional Acupuncture group.
  Interventions: Other: Acupuncture
- Placebo Acupuncture (Placebo Comparator): Placebo needles designed by Streitberger (1998) will be used. The placebo needles are blunt needle that will not penetrate the skin during needle insertion. The handles of these placebo needles will slide over the needle when it is compressed, giving it the appearance of penetrating the skin. The placebo needles are inserted to the site 1 inch beside the acupoints in order to avoid the acupressure effect. The needles are held by a surgical tape or hair pin in hairy region to imitate the retention of needles. The needles are connected to an electric-stimulator with zero frequency and amplitude. The number, duration and frequency of the treatment sessions, and the intervention procedure will be the same for electro-acupuncture and placebo acupuncture.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture at bilateral Ear Shenmen, Sishencong EX-HN1, Anmian, and unilateral Yintang EX-HN3 and Baihui GV20. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Other Names: Electroacupuncture

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of acupuncture treatment on residual insomnia in major depressive patients.

DETAILED DESCRIPTION:
This is a randomized single-blinded controlled trial. Patients will be randomly assigned to one of the three groups. One is the traditional acupuncture treatment group, one is the non-traditional acupuncture treatment group and the other is an acupuncture-like placebo treatment. Patients will be put into groups and then compared. The chance of getting into each group is 1:1:1, i.e. equal chance.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give informed consent;
* Hong Kong resident;
* Age 18-65 years;
* Previous DSM-IV Major Depressive Disorder as confirmed with the Structured Clinical Interview for DSM-IV;
* Hamilton Depression Rating Scale scores of 18 or below for at screening and baseline visit;
* A chief complaint of insomnia;
* Able to comply with the trial protocol.

Exclusion Criteria:

* Any symptoms suggestive of specific sleep disorders, including loud snoring, periodic leg movement, parasomnia;
* A diagnosis of sleep apnea or periodic limb movement disorder (PLMD) as assessed by overnight polysomnography (PSG);
* Presence of suicidal risk;
* Previous history of schizophrenia, other psychotic disorders, and bipolar disorder;
* Pregnant, breast-feeding, or woman of childbearing potential not using adequate contraception;
* Infection or abscess close to the site of selected acupoints and in the investigator's opinion inclusion is unsafe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Self-rated sleep quality score measured by Insomnia Severity Index questionnaire | Baseline, weekly during the treatment course, 1-week and 4-week posttreatment.
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by objective measure - wrist actigraphy | Baseline, 1-week posttreatment, and 4-week posttreatment.
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by subjective measures using sleep log. | Baseline, weekly during the treatment course, 1-week and 4-week posttreatment.

SECONDARY OUTCOMES:
Self-rated sleep quality score measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Baseline, weekly during the treatment course, 1-week and 4-week posttreatment.
Depression state measured by Hamilton Depression Rating Scale (HAMD) | Baseline, 1-week posttreatment, and 4-week posttreatment.
Subjects' functioning regarding work/study, social life and family measured by Sheehan Disability Scale | Baseline, weekly during the treatment course, 1-week and 4-week posttreatment.
Subjects' credibility to the treatment measured by Credibility of treatment rating scale | Second and the last time of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Fai Chung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Western Psychiatry Centre, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Chung KF, Yu YB, Lao L. What predicts a positive response to acupuncture? A secondary analysis of three randomised controlled trials of insomnia. Acupunct Med. 2017 Mar;35(1):24-29. doi: 10.1136/acupmed-2016-011058. Epub 2016 Aug 8. PMID 27503746
- [Derived] Yeung WF, Chung KF, Tso KC, Zhang SP, Zhang ZJ, Ho LM. Electroacupuncture for residual insomnia associated with major depressive disorder: a randomized controlled trial. Sleep. 2011 Jun 1;34(6):807-15. doi: 10.5665/SLEEP.1056. PMID 21629370